CLINICAL TRIAL: NCT05415761
Title: Comparative Effectiveness of Mobile Health Smoking Cessation Approaches Among Underserved Patients in Primary Care
Acronym: PROMOTE-UP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202200918; OCR41824 (Other: UF OnCore)
Record Dates: First submitted 2022-06-08; First posted 2022-06-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Tobacco Use Cessation
Keywords: tobacco use intervention; mobile health aids
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized to one of the 3 study arms, using a 1:1:1 allocation scheme
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iCanQuit (Active Comparator): iCanQuit is a modern, cognitive behavioral treatment which promotes cessation through greater acceptance of triggers for smoking and commitment to personal values. It is a smart phone-based acceptance and commitment therapy (ACT). For patients randomized to the iCanQuit arm (444 total), research staff will assist in downloading the app onto the patient's phone.
  Interventions: Behavioral: iCanQuit
- iCanQuit+Motiv8 (Active Comparator): Motiv8 is an internet-and smart phone-based contingency management (CM) intervention. Motiv8 verifies smoking status via a hand-held breath carbon monoxide (CO) monitor that is connected to a smart phone. For patients randomized to the iCanQuit+Motiv8 arm (444 total), research staff will assist in downloading the combined pp and connecting the iCO to the patient's phone. Smokers will also be asked to complete the first 4 iCanQuit modules, which contain exercises designed to prepare the users for their quit day. The end of the preparation phase will also mark each patient's quit date. During the intervention (7 weeks), participants will be considered abstinent from smoking if their breath CO sample is ≤ 5 ppm or if the CO value has decreased by 5% per hour from the last sample provided.
  Interventions: Behavioral: iCanQuit+Motiv8
- Florida quit line (Active Comparator): The Florida quit line provides telephone counseling for smoking cessation. Patients randomized to the Florida quit line arm (444 total) will be enrolled after contact information is sent electronically.
  Interventions: Behavioral: Florida quit line

INTERVENTIONS:
Behavioral: iCanQuit — iCanQuit is a smoking cessation smart phone application that uses acceptance and commitment therapy (ACT) approach, a cognitive behavioral treatment
  Arms: iCanQuit
Behavioral: iCanQuit+Motiv8 — iCanQuit + Motiv8 is a integrated version of iCanQuit (Cognitive Behavioral Therapy smoking cessation therapy application) with Motiv8 (a contingency management program that rewards decreased smoking determined by measuring CO levels of participant)
  Arms: iCanQuit+Motiv8
Behavioral: Florida quit line — An evidence-based, existing smoking cessation healthcare option recommended by the U.S. clinical practice that connects active smokers to trained quit coaches via referral by their providers.
  Arms: Florida quit line

SUMMARY:
This study will evaluate the comparative effectiveness of three smoking cessation therapies: mobile health (mHealth) application iCanQuit, mHealth application iCanQuit + Motiv8, and the Florida quit line.

DETAILED DESCRIPTION:
The research team will recruit 1,332 adult patients who smoke from primary care clinics in North Central Florida, focusing on: (a) the relative effectiveness of the 3 treatments in adult patients who smoke cigarettes, in underserved urban and rural primary care settings. The team will assign patients by chance to one of the 3 treatments. Smoking cessation will be confirmed with a breath test (measured at 2, 6, and 12 months). The study will measure the effects of these treatments in based on gender, race, ethnicity, rurality, and social vulnerability; (b) their effects on patients' quality of life, self-confidence in quitting, and satisfaction with the treatments; and (c) their impact on patients' reported levels of motivation, commitment to values, and acceptance of triggers for smoking.

ELIGIBILITY:
Inclusion Criteria:

* ≥21 years old
* Referred by the provider via Ask-Advise-Connect
* Receiving care at one of the participating clinics
* Daily access to their own smart phone (the study team will provide assistance to patients without a phone to obtain one through aid programs for low-income patients)
* No household members already enrolled

Exclusion Criteria:

* Unstable medical or psychiatric illness

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1332 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Smoking Point-Prevalence Abstinence (PPA) | Month 6
  negative CO breath sample ≤ 5 ppm using an iCO monitor, and self-reported abstinence from smoking in the last 7 days

SECONDARY OUTCOMES:
Smoking Point-Prevalence Abstinence (PPA) | Months 2 and 12
  negative CO breath sample ≤ 5 ppm using an iCO monitor, and self-reported abstinence from smoking in the last 7 days
Treatment Satisfaction | Month 12
  5-item scale measuring treatment by interest, usefulness, concern with privacy, how easy to understand, and satisfaction. Items will be measured on a 0-10 point scale, with higher scores corresponding to greater acceptability.
Quality of Life and Well-Being | Baseline, and month 6
  World Health Organization Quality of Life-BREF (WHOQOL-BREF): 26-item scale that measures quality of life. Items are rated on a 5-point Likert scale (low score of 1 to high score of 5), with a higher score indicating a higher quality of life.
Self Efficacy | Baseline, and month 6
  Self-Efficacy Questionnaire (SEQ-12): 12-item scale. Items are rated on a 5-point Likert scale (low score of 1 to high score of 5), with higher scores indicating greater self-efficacy.
Acceptance | Months 2 and 6
  9-item physical sensations subscale of the Avoidance and Inflexibility Scale. Items are rated on a 5-point Likert scale (low score of 1 to high score of 5), with higher scores reflecting more inflexibility/avoidance in the presence of difficult smoking-related thoughts, feelings, and sensations.
Values | Months 2 and 6
  Valuing Questionnaire (VQ): 10-item measure assessing the extent to which one lives consistently with their values, including Progress and Obstruction subscales. Both subscales total scores range from 0 to 30. A psychologically healthier score is indicated by a higher score on the Progress scale along with a lower score on the Obstructions scale.
Motivation | Months 2 and 6
  Motivational Engagement Questionnaire: 5-item measure. Items are rated on a 7-point Likert scale (low score of 1 to high score of 7), with higher scores indicating more motivation to quit smoking.
Smoking Prolonged Abstinence | Months 6 and 12
  Self-reported abstinence from the date of the last time a cigarette was smoked.

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Dallery, PhD, Principal Investigator — University of Florida; Ramzi Salloum, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Salloum RG, Bricker JB, Lee JH, Theis RP, Pluta K, Williams MP, Naous J, Mulani SR, Cogle CR, Rubin DA, Fahnlander AM, Nordelo B, Sullivan BM, Bloodworth S, Corbin L, Siler K, Willis D, Carrasquillo O, Dallery J. Comparative effectiveness of mobile health smoking cessation approaches among underserved patients in primary care: Study protocol for the PROMOTE-UP trial. Contemp Clin Trials. 2023 Apr;127:107120. doi: 10.1016/j.cct.2023.107120. Epub 2023 Feb 16. PMID 36804046